CLINICAL TRIAL: NCT06029114
Title: Magnetic Resonance Elastography of Cognitive Impairment
Brief Title: MR Elastography of Cognitive Impairment
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John Huston, Principal Investigator, Mayo Clinic
Other Study IDs: 23-004125; R01AG076636 (NIH)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Healthy
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control Group: Subjects will have a magnetic resonance elastography (MRE) performed.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography (MRE)
- Alzheimer's Disease Group: Subjects will have a magnetic resonance elastography (MRE) performed.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography (MRE)
- Mild Cognitive Impairment Group: Subjects will have a magnetic resonance elastography (MRE) performed.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography (MRE)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography (MRE) — Imaging technique performed on a Compact 3T MRI scanner that measures the stiffness (mechanical properties) of tissues.

SUMMARY:
The purpose of this research is to further investigate the potential of brain stiffness as a novel biomarker for Alzheimer's disease.

DETAILED DESCRIPTION:
Due to shifting demographics, the prevalence of dementia continues to increase in the population. To mitigate the effects of dementia will require new treatments working jointly with new methods for earlier and more sensitive diagnosis of the diseases. Magnetic resonance elastography (MRE) is a noninvasive technique for measuring tissue stiffness. MRE is a three-step process beginning with the introduction of shear waves into the tissue of interest with an external vibration source. The shear waves are imaged with a phase-contrast MRI pulse sequence and the resulting wave images are mathematically inverted to calculate tissue stiffness.

Preliminary data indicate that global brain stiffness is highly reproducible and that Alzheimer's disease causes a decrease in brain stiffness when compared to age- and gender-matched cognitively normal controls. The purpose of the proposed work is to further investigate the potential of brain stiffness as a novel biomarker for Alzheimer's disease. A comparison between brain stiffness and existing Alzheimer's disease biomarkers will help determine the biological basis of the observed stiffness change and in time may improve the sensitivity of Alzheimer's disease diagnosis and grading.

ELIGIBILITY:
Inclusion Criteria for Control Subjects:

* In good general health
* No Active neurological or psychiatric conditions, if a prior neurological or psychiatric condition was present they must have returned to normal
* No cognitive complaints
* Normal neurological examination
* No psychoactive medications
* They may have a chronic medical condition that does not affect cognition
* Low Aβ load Pittsburgh compound-B (PiB) ratio <1.5

Inclusion Criteria for Mild Cognitive Impairment Subjects:

* In good general health
* Memory complaint documented by the patient and collateral source
* Normal general cognitive function as determined by measure of general intellectual function and screening including the Short Test of Mental Status
* Normal activities of daily living as documented by history and Record of Independent Living
* Not demented by DSM-III-R criteria
* Do have an objective memory impairment determined by the clinical judgement of the neuropsychologists and neurologists
* High Aβ load Pittsburgh compound-B (PiB) ratio ≥1.5

Inclusion Criteria for Alzheimer's Disease Subjects:

* In good general health
* Dementia not a result of other medical or psychiatric conditions
* Diagnosis of dementia made according to DSM-III-R criteria
* Do have objective memory impairment determined by the clinical judgement of the neuropsychologists and neurologists
* High Aβ load Pittsburgh compound-B (PiB) ratio ≥1.5

Exclusion Criteria:

* Alzheimer's disease or mild cognitive impairment due to a known genetic mutation
* Major depression
* History of primary or metastatic intracranial neoplasm, significant head trauma, intra-cerebral hemorrhage, hemispheric stroke
* Contradictions to MRI imaging including but not limited to cardiac pacemakers, intraocular or intracranial metal, or other MRI incompatible devices.
* Pregnant women. Women of child bearing potential will be given a urine pregnancy test prior the MRI scan. Results will be shared with the participant. If the pregnancy test is positive, the participant will not be included within the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from Mayo Alzheimer's Disease Research Center.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Shear Stiffness | Baseline
  Brain stiffness measured by the magnetic resonance elastography (MRE) reported in Kilopascal (kPa)

SECONDARY OUTCOMES:
Joint mechanical-diffusion | Baseline
  MRE-based measurement of white matter regions of the brain

CONTACTS AND LOCATIONS:
Overall Officials: John Huston, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials